CLINICAL TRIAL: NCT04193098
Title: Phase I Clinical Study of Autologous Cytotoxic T Lymphocyte (CTL) Cell Immunotherapy Combination With PD-1 Inhibitor in the Second-line Treatment of Stage IIIB/IIIC/IV Non-Small Cell Lung Cancer
Brief Title: Study of Autologous Cytotoxic T Lymphocyte Immunotherapy Combination With PD-1 Inhibitor in the Advanced NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2019090A
Record Dates: First submitted 2019-12-08; First posted 2019-12-10 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Non-small Cell Lung Cancer; Second-line Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm: CTL plus PD-1 inhibitor (Experimental): CTL , Toripalimab Toripalimab intravenous infusion 240mg d1; CTL, 1x10^9, intravenous infusion,d14; Q3W.
  Interventions: Biological: CTL; Biological: Toripalimab

INTERVENTIONS:
Biological: CTL — CTL injection
  Other Names: Autologous cytotoxic T lymphocyte
Biological: Toripalimab — Toripalimab injection

SUMMARY:
This prospective, unicentric, open-labe phase I study is to evaluate the safety and effect of autologous cytotoxic T lymphocyte immunotherapy combination with PD-1 inhibitor in the second-line treatment of stage IIIB/IIIC/IV non-small cell lung cancer.

DETAILED DESCRIPTION:
In the stage IIIB/IIIC/IV NSCLC, patients received Toripalimab Injection (PD-1 inhibitor) 240mg, d1; CTL cells venous re-transfusion >=1x10^9, d14; Q3W; till disease progresion, or intolerable adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

Subjects who must meet all the following criteria should be selected:

1. Agreeing to participate in this study and signing a written informed consent.
2. Male or female,from 18 to 75 years (including 18 and 75 years).
3. The life expectancy will be longer than 3 months and can be followed up.
4. Patients with stage IIIB/IIIC/IV NSCLC were confirmed by histological /cytological and imaging examinations. According to RECIST 1.1 standard, there will be at least one measurable lesion.
5. Initial medical treatment.Patients with adenocarcinoma need wild type of EGFR gene and ALK fusion gene negative to be included in this study.
6. ECOG score will be 0 or 1 within 7 days before randomization.
7. Within 14 days before the start of treatment, the results of laboratory test of blood routine, liver, kidney function and hormone levels must be met the following criteria:

   White blood cells: more than 3.0 × 109/L; Platelets: more than 100 × 109/L; Neutrophils: more than 1.5 × 109/L; Hemoglobin: more than 80g/L; Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN); Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN; Serum bilirubin: less than 1.25 × ULN; Serum creatinine: less than 1.25 × ULN. Cortisol and thyroid function will be in the normal range.
8. The toxicity and side effects of previous chemotherapy will must be alleviated to grade 1 or below (except hair loss).
9. Female subjects must take effective contraceptive measures throughout the study period; serum or urine pregnancy test results must be negative during screening and the whole study period.
10. Male subjects should take effective contraceptive measures from the beginning of treatment to within 6 months after the end of treatment.

Exclusion Criteria:

Subjects who meet any of the following criteria could not participate in this study:

1. Adenocarcinoma subjects with EGFR sensitive mutation or ALK translocation; molecular detection of EGFR-sensitive mutations or ALK translocations is not required in squamous carcinoma patients.
2. NSCLC that had received chemotherapy in the past.
3. Other malignant tumors needed treatment within five years.
4. Allogeneic tissue/organ transplantation.
5. Participating in research drug therapy within 4 weeks before the first administration of the trial.
6. Systemic glucocorticoid therapy or any other form of immunosuppressive therapy (except glucocorticoid preconditioned with docetaxel) is being administered within 3 days before the first administration of the experimental therapy.
7. Received anti-tumor monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy or major surgery within 4 weeks before the first use of the drug; received chest radiotherapy greater than 30 Gy within 6 months before the first use of the drug; and received chest radiotherapy with 30 Gy or less within 1 month before the first use of the drug.
8. Previous treatment with PD-1/PD-L1 antibodies.
9. Over the past two years, patients with active autoimmune diseases requiring systemic treatment, such as the use of corticosteroids, or immunosuppressants. Substitution therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction) is not a systemic treatment.
10. Patients with congenital or acquired immunodeficiency (e.g. HIV-infected persons), active hepatitis B (HBV-DNA > 10^3 copies/ml) or hepatitis C (hepatitis C antibody positive), and HCV-RNA higher than the detection limit of the analytical method.
11. Subjects with active central nervous system (CNS) metastases and/or cancerous meningitis.
12. Patients with active infections requiring systemic intravenous therapy. Mental illness or other illnesses, such as uncontrollable heart disease or pulmonary disease, diabetes, etc.
13. Subjects who are known to be allergic to any of the constituents of the drug being studied.
14. Subjects with a recent history of drug abuse (including alcohol) within one year.
15. Compliance is poor and can not cooperate with clinical research.
16. Female subjects who are pregnant or breastfeeding, or who are expected to be pregnant during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  ORR was calculated by the percentage of patients with a confirmed complete (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Xiubao Ren, M.D, Ph.D, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin